CLINICAL TRIAL: NCT05027529
Title: ECMOsorb Trial - Impact of a VA-ECMO in Combination With CytoSorb in Critically Ill Patients With Cardiogenic Shock- A Prospective, Randomized, Blinded, Monocenter Trial.
Brief Title: ECMOsorb Trial - Impact of a VA-ECMO in Combination With CytoSorb in Critically Ill Patients With Cardiogenic Shock
Acronym: ECMOsorb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Schulze (Other)
Responsible Party: Sponsor-Investigator, Christian Schulze, Prof. Dr. med., Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKSJ0131; DRKS00025265 (Registry Identifier: Deutsches Regsiter für Klinische Studien (DRKS))
Record Dates: First submitted 2021-03-12; First posted 2021-08-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock; VA-ECMO; venous arterial Extracorporeal Membrane Oxygenation; inotropic score; extracorporeal cytokine hemadsorption system; cytokine adsorber; intensive care; multi organ failure
MeSH Terms: conditions — Shock, Cardiogenic; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, blinded, monocenter trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: masking by using a "black-box"; the control group only receives a regular ECMO tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-ECMO and CytoSorb (Experimental): standard ICU care WITH CytoSorb
  Interventions: Device: CytoSorb
- VA-ECMO only (Placebo Comparator): standard ICU care WITHOUT CytoSorb
  Interventions: Other: VA-ECMO only

INTERVENTIONS:
Device: CytoSorb — An extracorporeal cytokine hemoadsorption system is integrated in the VA-ECMO circuit
  Other Names: Standard ICU care (with VA-ECMO) AND CytoSorb Adsorber
  Arms: VA-ECMO and CytoSorb
Other: VA-ECMO only — only VA-ECMO; NO extracorporeal cytokine hemoadsorption system is added
  Other Names: Standard ICU care (with VA-ECMO)
  Arms: VA-ECMO only

SUMMARY:
In the ECMOsorb study the impact of a veno-arterial -ECMO in combination with an extracorporeal cytokine hemadsorption system in critically ill patients with cardiogenic shock is to be examined

DETAILED DESCRIPTION:
The prospective, interventional, randomised controlled and blinded ECMOsorb study investigates in critically ill patinets with cardiogenic shock and with veno-arterial ECMO (VA-ECMO) treatment the impact of an extracorporeal cytokin hemadsorption system on hemodynamics, defined by the Inotropic Score 72 hours after initiation of the adsorber (intervention) or normal ECMO tube (control) in the VA-ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock of any cause and indication for VA-ECMO
* Age between 18 and 80
* Signed informed consent

Exclusion Criteria:

* Current participation in another interventional trial
* Pregnancy
* Current immunosuppressive or immunomodulatory therapy
* Contraindications to VA-ECMO implantation.
* Patients with pre - existing sepsis (raised CPR, positive PCT, leukozytosis, fever, positive blood cultures).
* Shock duration> 12 h before evaluation.
* Severe PVD (peripheral vessel disease) making ECMO-implantation impossible.
* Aortic valve insufficiency / stenosis at least II °.
* Age > 80 years.
* CNS disease with fixed, dilated pupils (not drug-induced).
* Severe concomitant disease with limited life expectancy <6 months.
* CPR> 60min.
* Shock due to other reasons
* HIT positive (Heparin induced thrombocytopenia)
* Very low platelet counts (< 20,000/µl)
* Body weight less than 45 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in inotropic score after 72h (difference between the two study groups) | 72 hours
  Inotropic Score: dopamine dose [μg/kg/min] + dobutamine dose [μg/kg/min] + 100x epinephrine dose [μg/kg/min] + 100x norepinephrine [μg/kg/min]

SECONDARY OUTCOMES:
Interleukin 6 | 0 to 7 days after beginning of intervention
  pg/ml
Procalcitonin | 0 to 7 days after beginning of intervention
  ng/ml
c-reactive protein | 0 to 7 days after beginning of intervention
  mg/l
lactate | 0 to 7 days after beginning of intervention
  mmol/l
creatinine | 0 to 7 days after beginning of intervention
  µmol/l
glomerular filtration rate (GFR) | 0 to 7 days after beginning of intervention
  ml/min
troponin | 0 to 7 days after beginning of intervention
  pg/ml
creatinine kinase | 0 to 7 days after beginning of intervention
  µmol/l*s
myoglobine | 0 to 7 days after beginning of intervention
  µg/l
urinary output | 0 to 7 days after beginning of intervention
  ml/h
neuron specific enolase | 0 to 7 days after beginning of intervention
  µg/l
s-100 | 0 to 7 days after beginning of intervention
  µg/l
cystatin c | 0 to 7 days after beginning of intervention
  mg/l
galectin-3 | 0 to 7 days after beginning of intervention
  ng/ml
Duration of: renal replacement therapy (CVVHD), mechanical ventilation, ECMO therapy, inotropic /vasopressor treatment | day 30 after beginning of intervention
  hours
30 day, ICU and in-hospital mortality | day 30 after beginning of intervention
  nominal scale (yes/no)
Length of stay in ICU and total length of hospital stay until discharge/transfer | day 30 after beginning of intervention
  hours
Necessary Implantation of an Active Assist Device or heart transplantation | day 30 after beginning of intervention
  nominal scale (yes/no)
SAPS II | 0 to 7 days after beginning of intervention
  Simplified Acute Physiology Score II (Minimum value: 0 / maximum value: 163; higher values means worse outcome)
APACHE II score | 0 to 7 days after beginning of intervention
  Acute Pysiology and Chronic Health Evaluation II (Minimum value: 0 / maximum value: 71; higher values means worse outcome)
SOFA score | 0 to 7 days after beginning of intervention
  Sequential Organ Failure Assessment Score (Minimum value: 0 / maximum value: 24; higher value means worse outcome)
cerebreal performance category (CPC) | 0 to 30 days after beginning of intervention
  CPC 1 (adequate function) to CPC 5 (brain dead)
Glasgow coma scale (GCS) | 0 to 30 days after beginning of intervention
  Assessment scheme for disorders of consciousness and brain function (eyes, verbal, motor); scale from 3 (severe impairment) to 15 points (no abnormalities)
EuroQuol 5D-3L Descriptive System | 7 to 30 days after beginning of intervention
  mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
EQ VAS | 7 to 30 days after beginning of intervention
  EQ visual analogue scale (EQ VAS), patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Modified Rankin scale | 0 to 30 days after beginning of intervention
  scale from 0 (no symptoms) to 6 (dead);
Measurement of right ventricular parameters | 0 to 7 days after beginning of intervention
  measurements of right ventricular function in the echo (TAPSE in mm; FAC in %; RVEDD in mm; sPAP in mmHg; RA area in cm²; TASV in cm/s; ICV in mm)
Measurement of left ventricular parameters | 0 to 7 days after beginning of intervention
  measurements of left ventricular function in the echo (LVEDD in mm; LVESD in mm; LVEF in %; VSD (yes/no); LVEDV in ml; LVESV in ml; GLS in %; LA volume in ml)
Measurement of kidney injury and kidney function | 0 to 7 days after beginning of intervention
  NGAL, KIM-1, L-FABP, IGFBP7 in ng/ml
Interleukin 18 | 0 to 7 days after beginning of intervention
  pg/ml
incidence of apoplexy | 30 days after beginning of intervention
  nominal scale (yes/no)
mean arterial pressure | 0 to 7 days after beginning of intervention
  mmHg
central venous oxygen saturation | 0 to 7 days after beginning of intervention
  in %
mixed venous oxygen saturation | 0 to 7 days after beginning of intervention
  in %
arterial oxygen saturation | 0 to 7 days after beginning of intervention
  in %
heart failure re-hospitalisation | 30 days after beginning of intervention
  nominal scale (yes/no)
Brain natriuretic peptide (BNP) | 0 to 7 days after beginning of intervention
  pg/ml
n-terminal pro brain natriuretic peptide (NT-proBNP) | 0 to 7 days after beginning of intervention
  pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schulze, Prof., Study Director — Jena University Hospital
Locations (1):
- Jena University Hospital, Department of Cardiology, Jena, Thuringia, Germany